CLINICAL TRIAL: NCT06601426
Title: NBI-NearFocus Assisted Cold Snare Polypectomy Improves the Complete Resection Rate of Small Colorectal Polyps: a Prospective Single-arm Observational Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xinyong Jia, chief physician, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 147258368
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colon Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NBI-NearFocus (Other): Narrow Band Imaging-NearFocus
  Interventions: Procedure: CSP

INTERVENTIONS:
Procedure: CSP — cold snare polypectomy

SUMMARY:
NBI-NearFocus can assist cold snare polypectomy (CSP) to remove small colorectal polyps, but its specific efficacy is not clear.The aim of this study was to assess the efficacy of CSP with NBI-NearFocus evaluation of polypectomy sites for removal of small colorectal polyps. And then formulate a standard operating procedure for cold snare removal of polyps.

ELIGIBILITY:
Inclusion Criteria:

① Outpatient or inpatient patients aged 18-85 years old;

② Untamed, subpodial, and flat polyps with a diameter of 5-9mm (Paris classification: O-Is O-Isp、O-IIa；JNET Classification: Typel, Type2A);

③ Patients who agree to participate in this study.

Exclusion Criteria:

* Individuals currently taking antiplatelet or anticoagulant drugs, or those with coagulation dysfunction (PT prolongation greater than 3 seconds);

  * Polyp diameter<5mm or ≥ 10mm, morphology does not conform or JNET classification ≥ Type 2B;

    * Individuals with severe heart, lung, liver and kidney dysfunction or severe mental disorders who cannot cooperate with the examination; ④ Patients with intestinal obstruction, inflammatory bowel disease, Lynch syndrome, and familial adenomatous polyposis diagnosis;

      * Pregnancy; ⑥ Those who fail to meet the requirements for bowel cleansing preparation (BBPS<6 points).

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Histopathological complete resection rate | 2-3 days

SECONDARY OUTCOMES:
Complete recovery rate of polyps | 2-3 days

CONTACTS AND LOCATIONS:
Overall Officials: Xinyong Jia, Principal Investigator — Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided